CLINICAL TRIAL: NCT06771986
Title: Soluble Advanced Glycation End Product (sRAGE) Levels in Childhood Obesity
Brief Title: Soluble Advanced Glycation End Product (sRAGE) Levels
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Pembe Soylu Ustkoyuncu, Principal investigator, Kayseri City Hospital
Other Study IDs: 791-2023
Record Dates: First submitted 2025-01-03; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Obese Patients
Keywords: Children, obesity, sRAGE
MeSH Terms: conditions — Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Other: Observation — sRAGE levels were studied in three different groups

SUMMARY:
The aim of this study is to evaluate sRAGE levels in children with obesity and to determine the relationship between metabolic status and sRAGE levels in childhood obesity

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Obesity BMI over 95th percentile BMI z-score over 2

Exclusion Criteria:

Primary hyperlipidemia Primary liver disease Hypothyroidism Diabetes

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese and Healthy children who admitted to Kayseri City Hospital
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of sRAGE levels in obese and healthy participants | From enrollment to the end of at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ustkoyuncu PS, Kocer D. Soluble receptor for advanced glycation end product (sRAGE) levels in adolescents with obesity, insulin resistance and metabolic syndrome: A case-control study and the review of the literature. BMC Endocr Disord. 2025 Sep 23;25(1):209. doi: 10.1186/s12902-025-02025-9. PMID 40983915